CLINICAL TRIAL: NCT01500629
Title: A Randomized, Double-Blind, Placebo-Controlled, Crossover Trial of a Topical Nasal Spray in the the Relief of Signs and Symptoms of an Acute Response to a Nasal Allergen Challenge
Brief Title: Study of a Topical Nasal Spray to Ease the Symptoms of Hayfever
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: McNeil Consumer Healthcare Division of McNEIL-PPC, Inc. (Industry)
Collaborators: Johnson & Johnson Consumer and Personal Products Worldwide (Industry)
Responsible Party: Sponsor
Organization: Johnson & Johnson Consumer and Personal Products Worldwide (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double
Other Study IDs: POCEXP0001
Record Dates: First submitted 2011-12-22; First posted 2011-12-28 (Estimated); Results first posted 2014-05-09 (Estimated); Last update posted 2017-02-27 (Actual); Status verified 2017-01

CONDITIONS: Rhinitis, Allergic, Seasonal
Keywords: Allergic Rhinitis; Hayfever; Pollen Allergy
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal; Rhinitis, Allergic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- C-1266-7 (Experimental): In a crossover design with subjects randomized to treatment sequence, each subject will receive 200 uL of device Intervention C-1266-7. After a washout period of approximately 14 days, subjects will receive 200 uL of device Intervention C-1266-6 (placebo).
  Interventions: Device: C-1266-7; Device: C-1266-6 (placebo)
- Placebo (Experimental): In a crossover design with subjects randomized to treatment sequence, each subject will receive 200 uL of device Intervention C-1266-6 (placebo). After a washout period of approximately 14 days, subjects will receive 200 uL of device Intervention C-1266-7.
  Interventions: Device: C-1266-7; Device: C-1266-6 (placebo)

INTERVENTIONS:
Device: C-1266-7 — Each subject will receive two sprays (50 uL per spray for a total of 100 uL) of Investigational Nasal Spray (C-1266-7) in each nostril, for a total of 200 uL per treatment.
  Other Names: Not yet marketed
Device: C-1266-6 (placebo) — Each subject will receive two sprays (50 uL per spray for a total of 100 uL) of Sham Nasal Spray (C-1266-6, placebo) in each nostril, for a total of 200 uL per treatment.
  Other Names: Not yet marketed

SUMMARY:
The purpose of this study is to see if a new nasal spray can reduce the signs and symptoms of allergic rhinitis (hayfever). Subjects' participation in the study will last approximately 4 to 6 weeks, and each of three study visits during that time will last a few hours. Subjects will be required to have several tests done including allergy and breathing tests. They will be exposed to the item they are allergic to and will have small paper discs put in their noses. Subjects will also have the inside of their noses examined and will be asked questions about the level of their allergy symptoms.

DETAILED DESCRIPTION:
This study is a randomized, double blind, placebo-controlled, 2-way cross over trial. Approximately 25 subjects with a history of seasonal grass and/or ragweed allergy symptoms will be enrolled in the study to ensure 20 complete the study.

Subjects will be randomized to one of two treatment sequences of experimental product (investigational nasal spray) and placebo (sham nasal spray). Subjects will be asymptomatic of nasal symptoms (i.e., sneezing, itchy nose, runny nose, and nasal congestion) for at least 2 weeks prior to screening, and at least 1 week after the latest use of concomitant medication for symptom control in order to be eligible to participate in this study. Any subject with a history of mild asthma will be required to undergo a Forced Expiratory Volume in 1 second (FEV1) test prior to each nasal challenge (diluent and allergen) throughout the study. Assessments will be completed pre- and post-diluent challenge and post-allergen challenge. The baseline assessment for symptom scores is defined as the assessment obtained after the diluent challenge but prior (-15 minutes prior to randomization) to the administration of the experimental product/sham control.

Using a 14-day wash out period (± 2days), subjects who continue to meet inclusion criteria will receive treatments according to their randomized sequence. Eligible allergic subjects will undergo nasal challenges with either grass or ragweed allergen outside their allergy season.

Severity of symptoms will be assessed by the subject on a scale of 0=no symptoms to 3=severe. Adverse events will be collected during each visit, as well as the day following each visit via telephone.

ELIGIBILITY:
Inclusion Criteria:

* History of grass and/or ragweed allergic rhinitis for at least 2 years prior to screening
* Positive skin test to grass and/or ragweed antigen within 12 months prior to screening
* Being asymptomatic of nasal symptoms (i.e., sneezing, itchy nose, runny nose, and nasal congestion) for at least 2 weeks prior to screening.
* Females of childbearing potential must be using a medically-acceptable method of birth control for at least one month prior to screening and agree to continue using it during participation in the study (abstinence is not an approved method).

Exclusion Criteria:

* Participation in another investigational therapy 30 days prior to screening
* Not willing to give informed consent
* Inability to understand the nature and requirements of the study, or to comply with the study procedures
* Use of antihistamines within 1 week prior to screening (or during study visits)
* History of respiratory disease other than allergic rhinitis, allergic conjunctivitis and mild asthma.
* Current smoker or recent ex-smoker defined as history of smoking or use of nicotine containing substances within 2 months prior to screening as determined by medical history or subjects verbal report.
* Other severe acute or chronic medical or psychiatric condition that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the Investigator, would make the subject inappropriate for entry into this study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2012-01; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel S Qi, MD, PhD, Study Director — McNeil Consumer Healthcare Division of McNEIL-PPC, Inc.
Locations (1):
- The University of Chicago, Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- C-1266-7 Then Placebo: In a crossover design with subjects randomized to treatment sequence, each subject will receive 200 uL of device Intervention C-1266-7. After a washout period of approximately 14 days, subjects will receive 200 uL of device Intervention C-1266-6 (placebo).
  C-1266-7: Each subject will receive two sprays (50 uL per spray for a total of 100 uL) of Investigational Nasal Spray (C-1266-7) in each nostril, for a total of 200 uL per treatment.
  Placebo: Each subject will receive two sprays (50 uL per spray for a total of 100 uL) of Sham Nasal Spray (C-1266-6, placebo) in each nostril, for a total of 200 uL per treatment.
- Placebo Then C-1266-7: In a crossover design with subjects randomized to treatment sequence, each subject will receive 200 uL of device Intervention C-1266-6 (placebo). After a washout period of approximately 14 days, subjects will receive 200 uL of device Intervention C-1266-7.
  C-1266-7: Each subject will receive two sprays (50 uL per spray for a total of 100 uL) of Investigational Nasal Spray (C-1266-7) in each nostril, for a total of 200 uL per treatment.
  Placebo: Each subject will receive two sprays (50 uL per spray for a total of 100 uL) of Sham Nasal Spray (C-1266-6, placebo) in each nostril, for a total of 200 uL per treatment.
Period: Period 1 (Single Dose)
Arm/Group | C-1266-7 Then Placebo | Placebo Then C-1266-7
Started | 11 | 10
Completed | 11 | 10
Not Completed | 0 | 0
Period: Washout Period of 14 to 30 Days
Arm/Group | C-1266-7 Then Placebo | Placebo Then C-1266-7
Started | 11 | 10
Completed | 10 | 10
Not Completed | 1 | 0
Not completed — Pregnancy | 1 | 0
Period: Period 2 (Single Dose)
Arm/Group | C-1266-7 Then Placebo | Placebo Then C-1266-7
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- C-1266-7: In a crossover design with subjects randomized to treatment sequence, each subject will receive 200 uL of device Intervention C-1266-7. After a washout period of approximately 14 days, subjects will receive 200 uL of device Intervention C-1266-6 (placebo).
  C-1266-7: Each subject will receive two sprays (50 uL per spray for a total of 100 uL) of Investigational Nasal Spray (C-1266-7) in each nostril, for a total of 200 uL per treatment.
  Placebo: Each subject will receive two sprays (50 uL per spray for a total of 100 uL) of Sham Nasal Spray (C-1266-6) in each nostril, for a total of 200 uL per treatment.
- Placebo: In a crossover design with subjects randomized to treatment sequence, each subject will receive 200 uL of device Intervention C-1266-6. After a washout period of approximately 14 days, subjects will receive 200 uL of device Intervention C-1266-7.
  C-1266-7: Each subject will receive two sprays (50 uL per spray for a total of 100 uL) of Investigational Nasal Spray (C-1266-7) in each nostril, for a total of 200 uL per treatment.
  Placebo: Each subject will receive two sprays (50 uL per spray for a total of 100 uL) of Sham Nasal Spray (C-1266-6) in each nostril, for a total of 200 uL per treatment.
- Total: Total of all reporting groups
Arm/Group | C-1266-7 | Placebo | Total
Number analyzed (Participants) | 11 | 10 | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.0 (5.64) | 31.6 (10.38) | 28.1 (8.71)
Gender [Count of Participants; unit: Participants]
  Female | 8 | 4 | 12
  Male | 3 | 6 | 9
Region of Enrollment [Number; unit: participants]
  United States | 11 | 10 | 21

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Total Nasal Symptom Score (TNSS) at 15 Minutes After the First Allergan Challenge
Description: The change from baseline in TNSS of sneezing, itchy nose, runny nose, and nasal congestion at 15 minutes after the first allergen challenge. TNSS was the sum of the severity of sneezing and the average score (left and right nostrils) for each of the following: itchy nose, runny nose, and nasal congestion. Severity of sneezing, itchy nose, runny nose, and nasal congestion were evaluated using a 4-point categorical scale where 0 = no symptoms, 1 = mild, 2 = moderate, 3 = severe. For the change from baseline in TNSS, the total possible minimum value is 0 (best) and the total possible maximum value is 12 (worst).
Time Frame: 15 minutes (±5 minutes)
Population: Analysis is based on the Intent-to-Treat (ITT) set, which included all randomized subjects.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | C-1266-7 | Placebo
Number analyzed (Participants) | 21 | 20
units on a scale | 2.90 (0.533) | 3.69 (0.542)
Statistical Analysis 1: Comparison: C-1266-7 vs Placebo; The following comparison was made: Allergen Block (C-1266-7) vs placebo. For this comparison, the following hypothesis was tested: Ho: µ1= µ2 against the two-sided alternative H1: µ1≠ µ2 where µ1 and µ2 are the mean values of the parameter variable for the two treatment groups; Test type: Superiority or Other; p = 0.156, Mixed Models Analysis; Treatment, period and sequence as fixed effects and subject as a random effect; Mean Difference (Final Values) = -0.79, 95% CI 2-sided [-1.90 to 0.33]

2. Secondary Outcome: Change From Baseline in the Total Nasal Symptom Score (TNSS) at 1 Hour After the First Allergen Challenge
Description: The change from baseline in TNSS of sneezing, itchy nose, runny nose, and nasal congestion at 1 hour after the first allergen challenge. TNSS was the sum of the severity of sneezing and the average score (left and right nostrils) for each of the following: itchy nose, runny nose, and nasal congestion. Severity of sneezing, itchy nose, runny nose, and nasal congestion were evaluated using a 4-point categorical scale where 0 = no symptoms, 1 = mild, 2 = moderate, 3 = severe. For the change from baseline in TNSS, the total possible minimum value is 0 (best) and the total possible maximum value is 12 (worst).
Time Frame: 1 hour
Population: Analysis is based on the Intent-to-Treat (ITT) set, which included all randomized subjects.
Measure: Mean (Standard Error); unit: units on a scale
Groups:
- Placebo: In a crossover design with subjects randomized to treatment sequence, each subject will receive 200 uL of device Intervention C-1266-6, (placebo). After a washout period of approximately 14 days, subjects will receive 200 uL of device Intervention C-1266-7.
  C-1266-7: Each subject will receive two sprays (50 uL per spray for a total of 100 uL) of Investigational Nasal Spray (C-1266-7) in each nostril, for a total of 200 uL per treatment.
  C-1266-6 (placebo): Each subject will receive two sprays (50 uL per spray for a total of 100 uL) of Sham Nasal Spray (C-1266-6, placebo) in each nostril, for a total of 200 uL per treatment.
Arm/Group | C-1266-7 | Placebo
Number analyzed (Participants) | 21 | 20
units on a scale | .98 (.0507) | 1.27 (.517)
Statistical Analysis 1: Comparison: C-1266-7 vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.625, Mixed Models Analysis; Treatment, period and sequence as fixed effects and subject as a random effect; Mean Difference (Final Values) = -0.28, 95% CI 2-sided [-1.49 to 0.92]

3. Secondary Outcome: Change From Baseline in the Total Nasal Symptom Score (TNSS) at 15 Minutes After the Second Allergen Challenge
Description: The change from baseline in TNSS of sneezing, itchy nose, runny nose, and nasal congestion at 15 minutes after the second allergen challenge. TNSS was the sum of the severity of sneezing and the average score (left and right nostrils) for each of the following: itchy nose, runny nose, and nasal congestion. Severity of sneezing, itchy nose, runny nose, and nasal congestion were evaluated using a 4-point categorical scale where 0 = no symptoms, 1 = mild, 2 = moderate, 3 = severe. For the change from baseline in TNSS, the total possible minimum value is 0 (best) and the total possible maximum value is 12 (worst).
Time Frame: 15 minutes
Population: Analysis is based on the Intent-to-Treat (ITT) set, which included all randomized subjects.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Placebo: In a crossover design with subjects randomized to treatment sequence, each subject will receive 200 uL of device Intervention C-1266-6 (placebo).. After a washout period of approximately 14 days, subjects will receive 200 uL of device Intervention C-1266-7.
  C-1266-7: Each subject will receive two sprays (50 uL per spray for a total of 100 uL) of Investigational Nasal Spray (C-1266-7) in each nostril, for a total of 200 uL per treatment.
  C-1266-6 (placebo).: Each subject will receive two sprays (50 uL per spray for a total of 100 uL) of Sham Nasal Spray (C-1266-6, placebo) in each nostril, for a total of 200 uL per treatment.
Arm/Group | C-1266-7 | Placebo
Number analyzed (Participants) | 21 | 20
units on a scale | 2.73 (0.588) | 3.45 (0.600)
Statistical Analysis 1: Comparison: C-1266-7 vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.291, Mixed Models Analysis; Treatment, period and sequence as fixed effects and subject as a random effect; Mean Difference (Final Values) = -0.72, 95% CI 2-sided [-2.12 to 0.67]

4. Secondary Outcome: Change From Baseline in the Total Nasal Symptom Score (TNSS) at 1 Hour After the Second Allergen Challenge
Description: The change from baseline in TNSS of sneezing, itchy nose, runny nose, and nasal congestion at 1 hour after the second allergen challenge. TNSS was the sum of the severity of sneezing and the average score (left and right nostrils) for each of the following: itchy nose, runny nose, and nasal congestion. Severity of sneezing, itchy nose, runny nose, and nasal congestion were evaluated using a 4-point categorical scale where 0 = no symptoms, 1 = mild, 2 = moderate, 3 = severe. For the change from baseline in TNSS, the total possible minimum value is 0 (best) and the total possible maximum value is 12 (worst).
Time Frame: Within 1 hour
Population: Analysis is based on the Intent-to-Treat (ITT) set, which included all randomized subjects.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | C-1266-7 | Placebo
Number analyzed (Participants) | 21 | 20
units on a scale | 1.42 (0.630) | 1.49 (0.639)
Statistical Analysis 1: Comparison: C-1266-7 vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.899, Mixed Models Analysis; Treatment, period and sequence as fixed effects and subject as a random effect; Mean Difference (Final Values) = -0.07, 95% CI 2-sided [-1.21 to 1.07]

5. Secondary Outcome: Change From Baseline in Number of Sneezes at 15 Minutes After the First Allergen Challenge
Description: Change from baseline in number of sneezes
Time Frame: Within 15 minutes
Population: Analysis is based on the Intent-to-Treat (ITT) set, which included all randomized subjects.
Measure: Mean (Standard Deviation); unit: sneezes
Arm/Group | C-1266-7 | Placebo
Number analyzed (Participants) | 21 | 20
sneezes | 2.7 (4.22) | 2.1 (2.86)
Statistical Analysis 1: Comparison: C-1266-7 vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.701, Wilcoxon (Mann-Whitney) — The rank sum test was based on period difference for comparison between sequence; Median Difference (Final Values) = 0.0

6. Secondary Outcome: Change From Baseline in Number of Sneezes at 1 Hour After the First Allergen Challenge
Description: Change from baseline in number of sneezes
Time Frame: Within 1 hour
Population: Analysis is based on the Intent-to-Treat (ITT) set, which included all randomized subjects.
Measure: Mean (Standard Deviation); unit: sneezes
Arm/Group | C-1266-7 | Placebo
Number analyzed (Participants) | 21 | 20
sneezes | 0.0 (0.71) | 0.2 (1.61)
Statistical Analysis 1: Comparison: C-1266-7 vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.108, Wilcoxon (Mann-Whitney) — The rank sum test was based on period difference for comparison between sequence; Median Difference (Final Values) = 0.0

7. Secondary Outcome: Change From Baseline in Number of Sneezes at 15 Minutes After the Second Allergen Challenge
Description: Change from baseline in number of sneezes
Time Frame: Within 15 minutes
Population: Analysis is based on the Intent-to-Treat (ITT) set, which included all randomized subjects.
Measure: Mean (Standard Deviation); unit: sneezes
Arm/Group | C-1266-7 | Placebo
Number analyzed (Participants) | 21 | 20
sneezes | 1.1 (2.43) | 1.2 (1.18)
Statistical Analysis 1: Comparison: C-1266-7 vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.253, Wilcoxon (Mann-Whitney) — The rank sum test was based on period difference for comparison between sequence; Median Difference (Final Values) = -1.0

8. Secondary Outcome: Change From Baseline in Number of Sneezes at 1 Hour After the Second Allergen Challenge
Description: Change from baseline in number of sneezes
Time Frame: Within 1 hour
Population: Analysis is based on the Intent-to-Treat (ITT) set, which included all randomized subjects.
Measure: Mean (Standard Deviation); unit: sneezes
Groups:
- C-1266-7: In a crossover design with subjects randomized to treatment sequence, each subject will receive 200 uL of device Intervention C-1266-7. After a washout period of approximately 14 days, subjects will receive 200 uL of device Intervention C-1266-6.
  C-1266-7: Each subject will receive two sprays (50 uL per spray for a total of 100 uL) of Investigational Nasal Spray (C-1266-7) in each nostril, for a total of 200 uL per treatment.
  Placebo: Each subject will receive two sprays (50 uL per spray for a total of 100 uL) of Sham Nasal Spray (C-1266-6) in each nostril, for a total of 200 uL per treatment.
- Placebo: In a crossover design with subjects randomized to treatment sequence, each subject will receive 200 uL of device Intervention C-1266-6 (placebo). After a washout period of approximately 14 days, subjects will receive 200 uL of device Intervention C-1266-7.
  C-1266-7: Each subject will receive two sprays (50 uL per spray for a total of 100 uL) of Investigational Nasal Spray (C-1266-7) in each nostril, for a total of 200 uL per treatment.
  Placebo: Each subject will receive two sprays (50 uL per spray for a total of 100 uL) of Sham Nasal Spray (C-1266-6) in each nostril, for a total of 200 uL per treatment.
Arm/Group | C-1266-7 | Placebo
Number analyzed (Participants) | 21 | 20
sneezes | 0.0 (0.80) | 0.1 (1.59)
Statistical Analysis 1: Comparison: C-1266-7 vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.287, Wilcoxon (Mann-Whitney) — The rank sum test was based on period difference for comparison between sequence; Median Difference (Final Values) = 0.0

9. Secondary Outcome: Change From Baseline of Individual Nasal Symptoms Score (NSS) for Sneezing at 15 Minutes After the First Allergen Challenge
Description: Subjects evaluated the individual nasal symptom of sneezing using a scale of 0 = no symptoms, 1 = mild, 2 = moderate, and 3 = severe. The change from baseline of the individual NSS for sneezing was then calculated by taking the score at the post baseline time point minus its baseline score. For the change from baseline in the individual NSS for sneezing, the total possible minimum value is 0 (best) and the total possible maximum value is 3 (worst).
Time Frame: Within 15 minutes
Population: Analysis is based on the Intent-to-Treat (ITT) set, which included all randomized subjects.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | C-1266-7 | Placebo
Number analyzed (Participants) | 21 | 20
units on a scale | 0.8 (1.41) | 1.1 (1.10)
Statistical Analysis 1: Comparison: C-1266-7 vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.409, Wilcoxon (Mann-Whitney) — The rank sum test was based on period difference for comparison between sequence; Median Difference (Final Values) = 0.0

10. Secondary Outcome: Change From Baseline of Individual Nasal Symptoms Score (NSS) for Sneezing at 1 Hour After the First Allergen Challenge
Description: as for outcome 9
Time Frame: Within 1 hour
Population: Analysis is based on the Intent-to-Treat (ITT) set, which included all randomized subjects.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | C-1266-7 | Placebo
Number analyzed (Participants) | 21 | 20
units on a scale | -0.1 (1.00) | 0.5 (1.05)
Statistical Analysis 1: Comparison: C-1266-7 vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.092, Wilcoxon (Mann-Whitney) — The rank sum test was based on period difference for comparison between sequence; Median Difference (Final Values) = 0.0

11. Secondary Outcome: Change From Baseline of Individual Nasal Symptoms Score (NSS) for Sneezing at 15 Minutes After the Second Allergen Challenge
Description: as for outcome 9
Time Frame: Within 15 minutes
Population: Analysis is based on the Intent-to-Treat (ITT) set, which included all randomized subjects.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | C-1266-7 | Placebo
Number analyzed (Participants) | 21 | 20
units on a scale | 0.3 (1.06) | 1.1 (1.10)
Statistical Analysis 1: Comparison: C-1266-7 vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.042, Wilcoxon (Mann-Whitney) — The rank sum test was based on period difference for comparison between sequence; Median Difference (Final Values) = -1.0

12. Secondary Outcome: Change From Baseline of Individual Nasal Symptoms Score (NSS) for Sneezing at 1 Hour After the Second Allergen Challenge
Description: as for outcome 9
Time Frame: within 1 hour
Population: Analysis is based on the Intent-to-Treat (ITT) set, which included all randomized subjects.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | C-1266-7 | Placebo
Number analyzed (Participants) | 21 | 20
units on a scale | -0.0 (1.12) | 0.3 (0.85)
Statistical Analysis 1: Comparison: C-1266-7 vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.307, Wilcoxon (Mann-Whitney) — The rank sum test was based on period difference for comparison between sequence; Median Difference (Final Values) = 0.0

13. Secondary Outcome: Change From Baseline of Individual Nasal Symptoms Score (NSS) for Itchy Nose at 15 Minutes After the First Allergen Challenge
Description: Subjects evaluated the individual nasal symptom of itchy nose using a scale of 0 = no symptoms, 1 = mild, 2 = moderate, and 3 = severe. The change from baseline of the individual NSS for itchy nose was then calculated by taking the average score of the left and right nostrils for each score from each post baseline time point minus its baseline score. For the change from baseline in the individual NSS for itchy nose, the total possible minimum value is 0 (best) and the total possible maximum value is 3 (worst).
Time Frame: within 15 minutes
Population: Analysis is based on the Intent-to-Treat (ITT) set, which included all randomized subjects.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | C-1266-7 | Placebo
Number analyzed (Participants) | 21 | 20
units on a scale | 0.4 (0.55) | 0.5 (0.58)
Statistical Analysis 1: Comparison: C-1266-7 vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.903, Wilcoxon (Mann-Whitney) — The rank sum test was based on period difference for comparison between sequence; Median Difference (Final Values) = -0.5

14. Secondary Outcome: Change From Baseline of Individual Nasal Symptoms Score (NSS) for Itchy Nose at 1 Hour After the First Allergen Challenge
Description: as for outcome 13
Time Frame: within 1 hour
Population: Analysis is based on the Intent-to-Treat (ITT) set, which included all randomized subjects.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | C-1266-7 | Placebo
Number analyzed (Participants) | 21 | 20
units on a scale | 0.2 (0.49) | 0.2 (0.59)
Statistical Analysis 1: Comparison: C-1266-7 vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.121, Wilcoxon (Mann-Whitney) — The rank sum test was based on period difference for comparison between sequence; Median Difference (Final Values) = 0.0

15. Secondary Outcome: Change From Baseline of Individual Nasal Symptoms Score (NSS) for Itchy Nose at 15 Minutes After the Second Allergen Challenge
Description: as for outcome 13
Time Frame: Within 15 minutes
Population: Analysis is based on the Intent-to-Treat (ITT) set, which included all randomized subjects.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | C-1266-7 | Placebo
Number analyzed (Participants) | 21 | 20
units on a scale | 0.5 (0.73) | 0.5 (0.70)
Statistical Analysis 1: Comparison: C-1266-7 vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.689, Wilcoxon (Mann-Whitney) — The rank sum test was based on period difference for comparison between sequence; Median Difference (Final Values) = -0.3

16. Secondary Outcome: Change From Baseline of Individual Nasal Symptoms Score (NSS) for Itchy Nose at 1 Hour After the Second Allergen Challenge
Description: as for outcome 13
Time Frame: Within 1 hour
Population: Analysis is based on the Intent-to-Treat (ITT) set, which included all randomized subjects.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | C-1266-7 | Placebo
Number analyzed (Participants) | 21 | 20
units on a scale | 0.4 (0.73) | 0.3 (0.66)
Statistical Analysis 1: Comparison: C-1266-7 vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.314, Wilcoxon (Mann-Whitney) — The rank sum test was based on period difference for comparison between sequence; Median Difference (Final Values) = 0.0

17. Secondary Outcome: Change From Baseline of Individual Nasal Symptoms Score (NSS) for Runny Nose at 15 Minutes After the First Allergen Challenge
Description: Subjects evaluated the individual nasal symptom of runny nose using a scale of 0 = no symptoms, 1 = mild, 2 = moderate, and 3 = severe. The change from baseline of the individual NSS for runny nose was then calculated by taking the average score of the left and right nostrils for each score from each post baseline time point minus its baseline score. For the change from baseline in the individual NSS for runny nose, the total possible minimum value is 0 (best) and the total possible maximum value is 3 (worst).
Time Frame: Within 15 minutes
Population: Analysis is based on the Intent-to-Treat (ITT) set, which included all randomized subjects.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | C-1266-7 | Placebo
Number analyzed (Participants) | 21 | 20
units on a scale | 0.8 (0.86) | 1.4 (0.89)
Statistical Analysis 1: Comparison: C-1266-7 vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.034, Wilcoxon (Mann-Whitney) — The rank sum test was based on period difference for comparison between sequence; Median Difference (Final Values) = -0.8

18. Secondary Outcome: Change From Baseline of Individual Nasal Symptoms Score (NSS) for Runny Nose at 1 Hour After the First Allergen Challenge
Description: as for outcome 17
Time Frame: within 1 hour
Population: Analysis is based on the Intent-to-Treat (ITT) set, which included all randomized subjects.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | C-1266-7 | Placebo
Number analyzed (Participants) | 21 | 20
units on a scale | 0.3 (0.77) | 0.3 (0.41)
Statistical Analysis 1: Comparison: C-1266-7 vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.845, Wilcoxon (Mann-Whitney) — The rank sum test was based on period difference for comparison between sequence; Median Difference (Final Values) = 0.0

19. Secondary Outcome: Change From Baseline of Individual Nasal Symptoms Score (NSS) for Runny Nose at 15 Minutes After the Second Allergen Challenge
Description: as for outcome 17
Time Frame: within 15 minutes
Population: Analysis is based on the Intent-to-Treat (ITT) set, which included all randomized subjects.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | C-1266-7 | Placebo
Number analyzed (Participants) | 21 | 20
units on a scale | 1.0 (1.00) | 1.1 (0.90)
Statistical Analysis 1: Comparison: C-1266-7 vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.619, Wilcoxon (Mann-Whitney) — The rank sum test was based on period difference for comparison between sequence; Median Difference (Final Values) = 0.0

20. Secondary Outcome: Change From Baseline of Individual Nasal Symptoms Score (NSS) for Runny Nose at 1 Hour After the Second Allergen Challenge
Description: as for outcome 17
Time Frame: within 1 hour
Population: Analysis is based on the Intent-to-Treat (ITT) set, which included all randomized subjects.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | C-1266-7 | Placebo
Number analyzed (Participants) | 21 | 20
units on a scale | 0.5 (0.97) | 0.5 (0.85)
Statistical Analysis 1: Comparison: C-1266-7 vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.803, Wilcoxon (Mann-Whitney) — The rank sum test was based on period difference for comparison between sequence; Median Difference (Final Values) = 0.0

21. Secondary Outcome: Change From Baseline of Individual Nasal Symptoms Score (NSS) for Nasal Congestion at 15 Minutes After the First Allergen Challenge
Description: Subjects evaluated the individual nasal symptom of nasal congestion using a scale of 0 = no symptoms, 1 = mild, 2 = moderate, and 3 = severe. The change from baseline of the individual NSS for nasal congestion was then calculated by taking the average score of the left and right nostrils for each score from each post baseline time point minus its baseline score. For the change from baseline in the individual NSS for nasal congestion, the total possible minimum value is 0 (best) and the total possible maximum value is 3 (worst).
Time Frame: within 15 minutes
Population: Analysis is based on the Intent-to-Treat (ITT) set, which included all randomized subjects.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | C-1266-7 | Placebo
Number analyzed (Participants) | 21 | 20
units on a scale | 1.0 (0.72) | 0.8 (0.85)
Statistical Analysis 1: Comparison: C-1266-7 vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.175, Wilcoxon (Mann-Whitney) — The rank sum test was based on period difference for comparison between sequence; Median Difference (Final Values) = 0.3

22. Secondary Outcome: Change From Baseline of Individual Nasal Symptoms Score (NSS) for Nasal Congestion at 1 Hour After the First Allergen Challenge
Description: as for outcome 21
Time Frame: within 1 hour
Population: Analysis is based on the Intent-to-Treat (ITT) set, which included all randomized subjects.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | C-1266-7 | Placebo
Number analyzed (Participants) | 21 | 20
units on a scale | 0.6 (0.68) | 0.4 (0.61)
Statistical Analysis 1: Comparison: C-1266-7 vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.206, Wilcoxon (Mann-Whitney); The rank sum test was based on period difference for comparison between sequence; Median Difference (Final Values) = 0.5

23. Secondary Outcome: Change From Baseline of Individual Nasal Symptoms Score (NSS) for Nasal Congestion at 15 Minutes After the Second Allergen Challenge
Description: as for outcome 21
Time Frame: within 15 minutes
Population: Analysis is based on the Intent-to-Treat (ITT) set, which included all randomized subjects.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | C-1266-7 | Placebo
Number analyzed (Participants) | 21 | 20
units on a scale | 1.0 (0.97) | 0.8 (0.86)
Statistical Analysis 1: Comparison: C-1266-7 vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.072, Wilcoxon (Mann-Whitney) — The rank sum test was based on period difference for comparison between sequence; Median Difference (Final Values) = 0.5

24. Secondary Outcome: Change From Baseline of Individual Nasal Symptoms Score (NSS) for Nasal Congestion at 1 Hour After the Second Allergen Challenge
Description: as for outcome 21
Time Frame: within 1 hour
Population: Analysis is based on the Intent-to-Treat (ITT) set, which included all randomized subjects.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | C-1266-7 | Placebo
Number analyzed (Participants) | 21 | 20
units on a scale | 0.6 (0.95) | 0.5 (.097)
Statistical Analysis 1: Comparison: C-1266-7 vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = .0140, Wilcoxon (Mann-Whitney) — The rank sum test was based on period difference for comparison between sequence; Median Difference (Final Values) = 0.5

25. Secondary Outcome: Total Ocular Symptoms Score (TOSS) at 15 Minutes After the First Allergen Challenge
Description: Subjects evaluated ocular symptoms of itchy eyes, watery eyes, and redness of eyes using a scale of 0 = no symptoms, 1 = mild, 2 = moderate, and 3 = severe. The TOSS was calculated by taking the sum of each average score (left and right eyes) for itchy eyes, watery eyes, and redness of eyes. For the TOSS, the total possible minimum value is 0 (best) and the total possible maximum value is 9 (worst).
Time Frame: within 15 minutes
Population: Analysis is based on the Intent-to-Treat (ITT) set, which included all randomized subjects.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | C-1266-7 | Placebo
Number analyzed (Participants) | 21 | 20
units on a scale | 0.39 (0.176) | 0.40 (0.177)
Statistical Analysis 1: Comparison: C-1266-7 vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.907, Mixed Models Analysis; Treatment, period and sequence as fixed effects and subject as a random effect; Mean Difference (Final Values) = -0.01, 95% CI 2-sided [-0.24 to 0.22]

26. Secondary Outcome: Total Ocular Symptoms Score (TOSS) at 1 Hour After the First Allergen Challenge
Description: as for outcome 25
Time Frame: within 1 hour
Population: Analysis is based on the Intent-to-Treat (ITT) set, which included all randomized subjects.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | C-1266-7 | Placebo
Number analyzed (Participants) | 21 | 20
units on a scale | 0.13 (0.116) | 0.18 (0.118)
Statistical Analysis 1: Comparison: C-1266-7 vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.666, Mixed Models Analysis; Treatment, period and sequence as fixed effects and subject as a random effect; Mean Difference (Final Values) = -0.05, 95% CI 2-sided [-0.28 to 0.18]

27. Secondary Outcome: Total Ocular Symptoms Score (TOSS) at 15 Minutes After the Second Allergen Challenge
Description: as for outcome 25
Time Frame: within 15 minutes
Population: Analysis is based on the Intent-to-Treat (ITT) set, which included all randomized subjects.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | C-1266-7 | Placebo
Number analyzed (Participants) | 21 | 20
units on a scale | 0.33 (0.171) | 0.34 (0.173)
Statistical Analysis 1: Comparison: C-1266-7 vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.972, Mixed Models Analysis; Treatment, period and sequence as fixed effects and subject as a random effect; Mean Difference (Final Values) = -0.00, 95% CI 2-sided [-0.29 to 0.28]

28. Secondary Outcome: Total Ocular Symptoms Score (TOSS) at 1 Hour After the Second Allergen Challenge
Description: as for outcome 25
Time Frame: within 1 hour
Population: Analysis is based on the Intent-to-Treat (ITT) set, which included all randomized subjects.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | C-1266-7 | Placebo
Number analyzed (Participants) | 21 | 20
units on a scale | 0.24 (0.187) | 0.10 (0.191)
Statistical Analysis 1: Comparison: C-1266-7 vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.521, Mixed Models Analysis; Treatment, period and sequence as fixed effects and subject as a random effect; Mean Difference (Final Values) = 0.14, 95% CI 2-sided [-0.31 to 0.59]

29. Secondary Outcome: Change From Baseline of Non Nasal Symptoms Score (NNSS) at 15 Minutes After the First Allergen Challenge
Description: Subjects evaluated non nasal symptoms of itchy throat, ear, and palate using a scale of 0 = no symptoms, 1 = mild, 2 = moderate, and 3 = severe. The change from baseline of NNSS was calculated by taking the difference of the NNSS score for each post baseline time point minus its baseline. For the NNSS, the total possible minimum value is 0 (best) and the total possible maximum value is 3 (worst).
Time Frame: within 15 minutes
Population: Analysis is based on the Intent-to-Treat (ITT) set, which included all randomized subjects.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | C-1266-7 | Placebo
Number analyzed (Participants) | 21 | 20
units on a scale | 0.46 (0.170) | 0.35 (0.172)
Statistical Analysis 1: Comparison: C-1266-7 vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.376, Mixed Models Analysis; Treatment, period and sequence as fixed effects and subject as a random effect; Mean Difference (Final Values) = 0.12, 95% CI 2-sided [-0.15 to 0.39]

30. Secondary Outcome: Change From Baseline of Non Nasal Symptoms Score (NNSS) at 1 Hour After the First Allergen Challenge
Description: as for outcome 29
Time Frame: within 1 hour
Population: Analysis is based on the Intent-to-Treat (ITT) set, which included all randomized subjects.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | C-1266-7 | Placebo
Number analyzed (Participants) | 21 | 20
units on a scale | 0.38 (0.138) | 0.29 (0.140)
Statistical Analysis 1: Comparison: C-1266-7 vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.350, Mixed Models Analysis; Treatment, period and sequence as fixed effects and subject as a random effect; Mean Difference (Final Values) = 0.10, 95% CI 2-sided [-0.11 to 0.30]

31. Secondary Outcome: Change From Baseline of Non Nasal Symptoms Score (NNSS) at 15 Minutes After the Second Allergen Challenge
Description: as for outcome 29
Time Frame: within 15 minutes
Population: Analysis is based on the Intent-to-Treat (ITT) set, which included all randomized subjects.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | C-1266-7 | Placebo
Number analyzed (Participants) | 21 | 20
units on a scale | 0.42 (0.180) | 0.43 (0.183)
Statistical Analysis 1: Comparison: C-1266-7 vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.947, Mixed Models Analysis; Treatment, period and sequence as fixed effects and subject as a random effect; Mean Difference (Final Values) = -0.01, 95% CI 2-sided [-0.36 to 0.34]

32. Secondary Outcome: Change From Baseline of Non Nasal Symptoms Score (NNSS) at 1 Hour After the Second Allergen Challenge
Description: as for outcome 29
Time Frame: within 1 hour
Population: Analysis is based on the Intent-to-Treat (ITT) set, which included all randomized subjects.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | C-1266-7 | Placebo
Number analyzed (Participants) | 21 | 20
units on a scale | 0.33 (0.187) | 0.39 (0.188)
Statistical Analysis 1: Comparison: C-1266-7 vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.651, Mixed Models Analysis; Treatment, period and sequence as fixed effects and subject as a random effect; Mean Difference (Final Values) = -0.05, 95% CI 2-sided [-0.30 to 0.19]

33. Secondary Outcome: Within Subject Improvement From Placebo in TNSS (Responder) at 15 Minutes After the First Allergen Challenge
Description: A responder was defined as within subject improvement from placebo in TNSS with improvement from placebo based on the change from baseline for TNSS.
Time Frame: within 15 minutes
Measure: Number; unit: participants
Arm/Group | C-1266-7 | Placebo
Number analyzed (Participants) | 21 | 0
participants | 13 |

34. Secondary Outcome: Within Subject Improvement From Placebo in TNSS (Responder) at 1 Hour After the First Allergen Challenge
Description: as for outcome 33
Time Frame: within 1 hour
Population: Analysis is based on the Intent-to-Treat (ITT) set, which included all randomized subjects.
Measure: Number; unit: participants
Arm/Group | C-1266-7 | Placebo
Number analyzed (Participants) | 21 | 0
participants | 10 |

35. Secondary Outcome: Within Subject Improvement From Placebo in TNSS (Responder) at 15 Minutes After the Second Allergen Challenge
Description: as for outcome 33
Time Frame: within 15 minutes
Population: Analysis is based on the Intent-to-Treat (ITT) set, which included all randomized subjects.
Measure: Number; unit: participants
Arm/Group | C-1266-7 | Placebo
Number analyzed (Participants) | 21 | 0
participants | 10 |

36. Secondary Outcome: Within Subject Improvement From Placebo in TNSS (Responder) at 1 Hour After the Second Allergen Challenge
Description: as for outcome 33
Time Frame: within 1 hour
Population: Analysis is based on the Intent-to-Treat (ITT) set, which included all randomized subjects.
Measure: Number; unit: participants
Groups:
- C-1266-7 Then C-1266-6: In a crossover design with subjects randomized to treatment sequence, each subject will receive 200 uL of device Intervention C-1266-7. After a washout period of approximately 14 days, subjects will receive 200 uL of device Intervention C-1266-6.
  C-1266-7: Each subject will receive two sprays (50 uL per spray for a total of 100 uL) of Investigational Nasal Spray (C-1266-7) in each nostril, for a total of 200 uL per treatment.
  C-1266-6: Each subject will receive two sprays (50 uL per spray for a total of 100 uL) of Sham Nasal Spray (C-1266-6) in each nostril, for a total of 200 uL per treatment.
- C-1266-6 Then C-1266-7: In a crossover design with subjects randomized to treatment sequence, each subject will receive 200 uL of device Intervention C-1266-6. After a washout period of approximately 14 days, subjects will receive 200 uL of device Intervention C-1266-7.
  C-1266-7: Each subject will receive two sprays (50 uL per spray for a total of 100 uL) of Investigational Nasal Spray (C-1266-7) in each nostril, for a total of 200 uL per treatment.
  C-1266-6: Each subject will receive two sprays (50 uL per spray for a total of 100 uL) of Sham Nasal Spray (C-1266-6) in each nostril, for a total of 200 uL per treatment.
Arm/Group | C-1266-7 Then C-1266-6 | C-1266-6 Then C-1266-7
Number analyzed (Participants) | 21 | 0
participants | 6 |

37. Secondary Outcome: Change From Baseline of the Total Score From the Following Nasal Symptoms (TNSSX [Total Nasal Symptom Score Excluding Sneezing]): Itchy Nose, Runny Nose, Nasal Congestion at 15 Minutes After the First Allergen Challenge
Description: TNSSX was derived by taking the sum of the average score of left and right nostrils for itchy nose, runny nose, and nasal congestion. Change from baseline of TNSSX was TNSSX for each post baseline time point minus its baseline. For the change from baseline of TNSSX, the total possible minimum value is 0 (best) and the total possible maximum value is 9 (worst).
Time Frame: within 15 minutes
Population: Analysis is based on the Intent-to-Treat (ITT) set, which included all randomized subjects.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | C-1266-7 | Placebo
Number analyzed (Participants) | 21 | 20
units on a scale | 2.15 (0.376) | 2.61 (0.383)
Statistical Analysis 1: Comparison: C-1266-7 vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.261, Mixed Models Analysis; Treatment, period and sequence as fixed effects and subject as a random effect; Mean Difference (Final Values) = -0.46, 95% CI 2-sided [-1.30 to 0.38]

38. Secondary Outcome: Change From Baseline of the Total Score From the Following Nasal Symptoms (TNSSX [Total Nasal Symptom Score Excluding Sneezing]): Itchy Nose, Runny Nose, Nasal Congestion at 1 Hour After the First Allergen Challenge
Description: as for outcome 37
Time Frame: within 1 hour
Population: Analysis is based on the Intent-to-Treat (ITT) set, which included all randomized subjects.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | C-1266-7 | Placebo
Number analyzed (Participants) | 21 | 20
units on a scale | 1.08 (0.337) | 0.82 (0.344)
Statistical Analysis 1: Comparison: C-1266-7 vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.481, Mixed Models Analysis; Treatment, period and sequence as fixed effects and subject as a random effect; Mean Difference (Final Values) = 0.27, 95% CI 2-sided [-0.51 to 1.04]

39. Secondary Outcome: Change From Baseline of the Total Score From the Following Nasal Symptoms (TNSSX [Total Nasal Symptom Score Excluding Sneezing]): Itchy Nose, Runny Nose, Nasal Congestion at 15 Minutes After the Second Allergen Challenge
Description: as for outcome 37
Time Frame: within 15 minutes
Population: Analysis is based on the Intent-to-Treat (ITT) set, which included all randomized subjects.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | C-1266-7 | Placebo
Number analyzed (Participants) | 21 | 20
units on a scale | 2.41 (0.443) | 2.39 (0.450)
Statistical Analysis 1: Comparison: C-1266-7 vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.961, Mixed Models Analysis; Treatment, period and sequence as fixed effects and subject as a random effect; Mean Difference (Final Values) = 0.02, 95% CI 2-sided [-0.85 to 0.89]

40. Secondary Outcome: Change From Baseline of the Total Score From the Following Nasal Symptoms (TNSSX [Total Nasal Symptom Score Excluding Sneezing]): Itchy Nose, Runny Nose, Nasal Congestion at 1 Hour After the Second Allergen Challenge
Description: as for outcome 37
Time Frame: within 1 hour
Population: Analysis is based on the Intent-to-Treat (ITT) set, which included all randomized subjects.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | C-1266-7 | Placebo
Number analyzed (Participants) | 21 | 20
units on a scale | 1.47 (0.504) | 1.24 (0.510)
Statistical Analysis 1: Comparison: C-1266-7 vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.546, Mixed Models Analysis; Treatment, period and sequence as fixed effects and subject as a random effect; Mean Difference (Final Values) = 0.24, 95% CI 2-sided [-0.57 to 1.04]

ADVERSE EVENTS:
Time Frame: Up to 63 days (+30 days for Serious Adverse Events)
Description: The safety analysis set included all subjects who used at least one dose of investigational product/placebo.
Arm/Group | C-1266-7 | Placebo
Serious Adverse Events (participants affected / at risk) | 1/21 | 0/20
Other Adverse Events (participants affected / at risk) | 1/21 | 2/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | C-1266-7 (N=21) | Placebo (N=20)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | C-1266-7 (N=21) | Placebo (N=20)
Nasopharyngitis (Infections and infestations) | 0 | 1
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Pregnancy of Partner (Social circumstances) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor has the right to publish results without PI approval. PI has right to present and/or publish research results and related background information, but must provide publication to Sponsor in advance with at least 30 days for review. Sponsor confidential information cannot be submitted for publication without Sponsor's written consent. Sponsor cannot require changes or extend the embargo. If requested, the PI will withhold the publication for ≤60 days to allow for patent application.